CLINICAL TRIAL: NCT02342964
Title: Comparative Study of Different Non-invasive Measurement Methods of Hepatic Fibrosis in Cystic Fibrosis
Brief Title: Comparison of Non-invasive Measurement Methods of Hepatic Fibrosis in Cystic Fibrosis
Acronym: MUCO-FIBRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RCB-2013-A01579-36
Record Dates: First submitted 2014-11-06; First posted 2015-01-21 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; hepatic fibrosis; hepatic cirrhosis; non-invasive methods of measurement; hepatic elasticity
MeSH Terms: conditions — Cystic Fibrosis; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MUCO-FIBRO (Other): Measures of hepatic elasticity
  Interventions: Other: Measure of hepatic elasticity

INTERVENTIONS:
Other: Measure of hepatic elasticity — Measure of hepatic elasticity by four non-invasive methods:
  Fibroscan, Fibrotest, SWE, MRE.

SUMMARY:
Non-invasive methods of the quantification of fibrosis may help to assess the development of fibrosis at a specific moment of the evolution of the disease, in the order to decide the initiation of treatment with ursodeoxycholic acid which may slow the progression to hepatic cirrhosis:

* FibroTest,
* The ultrasound impulse elastography, Fibroscan (FS)
* Ultrasound Elastography by ShearWave (SWE)
* Magnetic resonance elastography (MRE). The purpose of this study is to assess the contribution of these methods in the diagnosis of hepatic fibrosis during the evolution of the cystic fibrosis.

DETAILED DESCRIPTION:
The incidence of hepatobiliary disease in cystic fibrosis in the first 10 years of life is 2.5 to 1.8 / 100 patient-years, significantly decreasing during the second decade; generally 30-40% of children develop hepatic disease before 12 years. However, the hepatobiliary damage varies in its clinical and histological expression. The typical histological appearance of the liver is the focal biliary cirrhosis (or fibrosis) characterized by a heterogeneous distribution of portal fibrosis in the liver.

Complications of cirrhosis are responsible for 2.5% of deaths in patients with cystic fibrosis and represent the second cause of death after lung disease if we exclude deaths secondary to lung transplantation.

The diagnosis of hepatic disease at an early stage of development and the assessment of the progression of fibrosis are so difficult in the absence of sensitive and specific non-invasive diagnostic tests.

Non-invasive assessment of hepatic fibrosis is an important topic of study in recent years, because of the emergence of biological methods and quantitative elastography methods using ultrasound or Magnetic Resonance Imagery (MRI) and allowing quantification of the hepatic elasticity, which is assumed to be a reflection of fibrosis. The advantages of these methods are numerous:

* The assessment of wider hepatic parenchyma then hepatic biopsy, allowing overcome the sampling bias
* Painless and non-invasive methods for the patient
* Simple to make
* Do not require hospitalization and can be performed as outpatient
* Immediately known results
* Can be repeated as often as necessary during the patient's follow-up
* Lower cost, morbidity and mortality compared to hepatic biopsy. Several non-invasive methods of fibrosis diagnosis have been studied in adults primarily for viral diseases and helped to limit the indications of hepatic biopsy. However, no method is now validated for the early diagnosis of hepatic disease and monitoring of children with cystic fibrosis.

The main objective of the study is to assess the contribution of FibroTest, the ultrasound impulse elastography, Fibroscan (FS), the ultrasound elastography by ShearWave (SWE) and Magnetic Resonance Elastography (MRE ) in the diagnosis of hepatic fibrosis in cystic fibrosis.

The secondary objectives are following :

* To study the correlations between the fibrosis quantitative results obtained through the four techniques of measurement and the matches between the results of four techniques using the standards available at t0 and after a year (t1).
* Study the correlations between clinical, biological and ultrasound endpoints of hepatic disease and various non-invasive measurement methods of fibrosis.
* Evaluate the area under the ROC curve of the different tests and the diagnostic performance tests using analytical methods without gold standard by classifying the children into two groups: the presence of advanced fibrosis (stages F2 to F4 ) or not (F0 and F1 stages), contracting by a committee according to the results of any biopsy, clinical, laboratory and ultrasound endpoints independent on the tests.

ELIGIBILITY:
Inclusion Criteria:

* Children with cystic fibrosis aged 6-18 years. The diagnosis of cystic fibrosis will be based on testing the abnormal sweat (> 60 mEq / L of chloride sweat) and / or on the presence of two pathogen mutations of CFTR.
* Written consent of parents or holders of parental rights.
* Affiliated or benefiting from a national social insurance

Exclusion Criteria:

* Presence of another disease associated with cystic fibrosis that may be responsible for a chronic hepatic disease such as deficiency of alpha-1antitrypsine ZZ genotype or chronic infection by virus B or C.
* Child grafted
* Actual febrile pulmonary infection that can change the value of Fibrotest
* Important peri-hepatic ascites preventing the elasticity measurements by Fibroscan®
* Severe respiratory insufficient preventing attainment of Magnetic Resonance Imagery

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Measure of hepatic elasticity by Fibro Test | Day 0
  The value of hepatic elasticity measured by each of the tests performed on the same day in the same patient
Measure of hepatic elasticity by the ultrasound impulse elastography, Fibroscan (FS) | Month 12
  The value of hepatic elasticity measured by each of the tests performed on the same day in the same patient.

SECONDARY OUTCOMES:
Measure of hepatic elasticity by Ultrasound Elastography by ShearWave (SWE): | Day 0
  The existence of advanced hepatic fibrosis (stages F2 to F4) will be defined by the presence of clinical, and / or biological and / or ultrasound abnormalities, defining two groups of children (F + :children with advanced fibrosis, F-: children with little or no fibrosis
Measure of hepatic elasticity by Magnetic resonance elastography (MRE): | Month 12
  The existence of advanced hepatic fibrosis (stages F2 to F4) will be defined by the presence of clinical, and / or biological and / or ultrasound abnormalities, defining two groups of children (F + :children with advanced fibrosis, F-: children with little or no fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Debray, MD, PhD, Principal Investigator — 00 33 1 44 49 41 52
Locations (1):
- Hôpital Necker, Paris, France

REFERENCES:
- [Result] Dana J, Girard M, Franchi-Abella S, Berteloot L, Benoit-Cherifi M, Imbert-Bismut F, Sermet-Gaudelus I, Debray D. Comparison of Transient Elastography, ShearWave Elastography, Magnetic Resonance Elastography and FibroTest as routine diagnostic markers for assessing liver fibrosis in children with Cystic Fibrosis. Clin Res Hepatol Gastroenterol. 2022 Mar;46(3):101855. doi: 10.1016/j.clinre.2021.101855. Epub 2021 Dec 20. PMID 34933150